CLINICAL TRIAL: NCT01892306
Title: Transdiagnostic Treatment for Anxiety and Bipolar I Disorder
Brief Title: Pilot Study of Cognitive Behavioral Therapy for Anxiety and Bipolar I Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Bipolar Clinic and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1F32MH098490-01 (NIH)
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Bipolar Disorder; Anxiety Disorders
MeSH Terms: conditions — Bipolar Disorder; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual plus UP CBT (Experimental): Existing psychiatrist-administered psychopharmacotherapy plus weekly transdiagnostic CBT
  Interventions: Behavioral: UP CBT
- Treatment as usual (Active Comparator): Existing psychiatrist-administered psychopharmacotherapy
  Interventions: Drug: Treatment as usual

INTERVENTIONS:
Behavioral: UP CBT — The UP is an 18-session weekly cognitive behavioral intervention for anxiety and mood disorders
  Other Names: Unified Protocol (UP) for transdiagnostic treatment of emotional disorders
  Arms: Treatment as usual plus UP CBT
Drug: Treatment as usual — Existing optimized pharmacotherapy as delivered by treating psychiatrist
  Arms: Treatment as usual

SUMMARY:
The specific goal of this research study is to investigate the feasibility, acceptability, and preliminary efficacy of a transdiagnostic, cognitive-behavioral therapy developed specifically to target common core processes across mood and anxiety disorders [Unified Protocol for Transdiagnostic Treatment of Emotional Disorders (UP)], for the treatment of patients with bipolar I disorder (BD-I) and comorbid anxiety. The study will compare treatment-as-usual with pharmacotherapy (TAU) plus 18 one-hour sessions of treatment with the UP to TAU alone. Patients in both treatment conditions will be followed over a 12-month period and will be assessed monthly to track changes in mood, anxiety and emotion-related symptoms; functional impairment; and relapse rates. Data on the acceptability of the treatment will be gathered concurrently through monthly patient self-reported ratings of treatment satisfaction, and by tracking rates of acceptance for randomization into the study, number of completed sessions, and dropout rates. The study will examine: 1) whether combined cognitive behavioral treatment (UP) for BD-I and comorbid anxiety disorders is an acceptable and feasible approach to treatment; 2) whether treatment with the UP for BD-I and comorbid anxiety disorders as an adjunct to pharmacotherapy treatment-as-usual (TAU) leads to greater symptom reduction and reduced functional impairment than pharmacotherapy alone, 3) whether treatment for BD-I and comorbid anxiety disorders with the UP improves relapse rates over a 6-month follow-up relative to TAU; and 4) whether reduction in symptoms, relapse rates, and functional impairment are mediated by changes in emotion regulation skills. The broader aim of this study is to address the need for improved treatments for bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65
* DSM-IV diagnosis of bipolar I disorder and at least one of three additional anxiety disorders:

generalized anxiety disorder, panic disorder, or social phobia.

* HAM-D-17 score <16 (i.e. depressive symptoms)
* YMRS score < 12 (i.e. no or very low manic symptoms)
* Current, stabilized (> 3 months) pharmacotherapy treatment under the care of a psychiatrist consisting of optimized, stable maintenance pharmacotherapy at maximum tolerated dosages according to Texas Implementation of Medication Algorithm.

Exclusion Criteria:

* Active suicidality (HAM-D-17 suicide item #3 score > 3) in the past 2 months. Potential participants scoring 3 or higher on the HAM-D-17 suicide item will be immediately evaluated by the PI and Sponsor and referred to a higher level of care if clinically indicated.
* DSM-IV bipolar I disorder subtype rapid cycling
* DSM-IV manic or mixed episode in the past 2 months
* DSM-IV major depressive episode in the past 2 months
* Psychotropic medication not in accordance with the revised Texas Implementation of Medication Algorithm
* Current Pregnancy
* Medical illness or non-psychiatric medical treatment that would likely interfere with study participation.
* Neurologic disorder, previous ECT, or history of head trauma (i.e. known structural brain lesion)
* Current or past history of selected DSM-IV Axis I disorders other than bipolar disorder including: organic mental disorder, substance abuse within the past 12 months and/or history of substance abuse for > 1 year; current substance dependence (including alcohol), as assessed by the Structured Clinical Interview for DSM-IV-TR, Substance Use Disorders (Section E); schizophrenia, delusional disorder, psychotic disorders not otherwise specified, obsessive compulsive disorder and posttraumatic stress disorder (due to low prevalence of ~6.5% each).
* Concurrent psychotherapy other than cognitive-behavioral therapy as provided in this study (to rule out other uncontrolled effects of concurrent psychotherapies)
* Presence of metallic implants that would interfere with safety during fMRI scanning (i.e. cardiac pacemaker, metal plates, etc.)
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital Bipolar Clinic and Research Program, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 were invited to consent. 34 consented to be screened for inclusion. 5 did not meet study inclusion criteria thus were not randomized (1 not on a stabilized medication; 1 did not meet criteria for anxiety disorder; 2 were currently substance dependent; 1 reported psychosis). 29 were randomized to TAU or TAU plus 18 sessions of CBT (UP+TAU).
Pre-assignment Details: Participants were excluded from the trial before assignment to study arms based on exclusion criteria related to diagnosis and unstable medication regime.
Period: Overall Study
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Started | 13 | 16
Completed | 8 | 10
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual | Total
Number analyzed (Participants) | 13 | 16 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.08 (13.84) | 44.25 (14.27) | 43.72 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Difficulties in Emotion Regulation Scale (DERS) [Mean (Standard Deviation); unit: units on a scale] — Emotion regulation skills were assessed at baseline using a self-report questionnaire measure of emotion regulation (Difficulties in Emotion Regulation Scale- DERS), a 36-item Likert-type scale (1-6) calculated by averaging scores across all items (minimum score 1, maximum score 6). Higher scores indicate greater impairment in emotion regulation skills.
  units on a scale | 2.84 (0.53) | 3.00 (0.56) | 2.92 (0.54)
Affective Control Scale (ACS) [Mean (Standard Deviation); unit: units on a scale] — Perceived controllability of emotions was assessed at baseline using the the self-report Affective Control Scale (ACS) a 42-item Likert-type scale (1-7) calculated by averaging scores across all items (minimum score 1, maximum score 7). Higher scores indicate greater impairment and less perceived control of emotions.
  units on a scale | 4.48 (0.70) | 4.24 (0.53) | 4.36 (0.61)
Anxiety Sensitivity Index (ASI) [Mean (Standard Deviation); unit: units on a scale] — Anxiety sensitivity was assessed at baseline using the self-report Anxiety Sensitivity Index questionnaire (ASI) a 16-item likert-type scale (0-4) calculated by summing scores across items (minimum score 0, maximum score 64). Higher scores indicate greater impairment.
  units on a scale | 33 (10.07) | 26.56 (13.47) | 29.45 (12.30)
NEO Five Factor Inventory of Personality, Neuroticism Subscale (NEO-FFI-N) [Mean (Standard Deviation); unit: units on a scale] — Neuroticism was assessed at baseline using the NEO Five Factor Personality Inventory Neuroticism Scale (NEO-FFI-N) which is a subscale of the NEO-FFI, a 60-item scale (0-4) calculated by summing scores for each subscale. Only the 12-item Neuroticism subscale is included in this study. Higher scores indicate greater impairment.
  units on a scale | 5.69 (1.03) | 5.88 (1.54) | 5.79 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: Reductions Over Time in Anxiety Symptoms as Measured by Hamilton Anxiety Rating Scale
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a well-validated clinician administered rating of anxiety-related symptoms. Ratings are made on a 0 (no symptoms) to 4 (most severe in frequency/duration/interference/distress) for each item (14 items), with a minimum score of 0 and a maximum score of 56 calculated by summing scores of all 14 items. Higher scores indicate greater impairment.
Time Frame: Six months
Population: ITT analysis, data imputed to account for 30% missing data. A total of 28 people were included in the ITT analysis - one TAU participant initiated CBT through a private practitioner mid-study (an exclusion criteria) and was subsequently excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
Units on scale
  Baseline | 14 (7.8) | 18.81 (6.10)
  Month 2 | 11.78 (8.99) | 17.70 (7.62)
  Month 3 | 13.86 (9.30) | 22.33 (7.68)
  Month 4 | 13.5 (7.03) | 18 (8.87)
  Month 5 | 10 (5.55) | 19.1 (8.29)
  Month 6 | 15.71 (10.29) | 18.89 (10.82)
Statistical Analysis 1: Comparison: Treatment as Usual Plus UP CBT; Scores on the HAM-A were analyzed using a mixed-effects linear regression analysis over 6 timepoints; Test type: Superiority or Other; p = .02, Mixed Models Analysis

2. Primary Outcome: Reductions Over Time in Depression Symptoms as Measured by Hamilton Depression Rating Scale (HAM-D)
Description: The Hamilton Depression Rating Scale (HAM-D) is a well-validated clinician administered rating of depression-related symptoms. Scores are calculated by summing scores across all 17-items, with a minimum score of 0 and a maximum score of 54. Higher scores indicate greater impairment.
Time Frame: Six months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
Units on scale
  Baseline | 10.54 (6.96) | 13.63 (4.87)
  Month 2 | 8 (7.94) | 11.2 (6.60)
  Month 3 | 11.86 (6.12) | 16.89 (6.13)
  Month 4 | 11.63 (6.63) | 11.9 (5.13)
  Month 5 | 9 (6.36) | 16 (5.70)
  Month 6 | 10.14 (7.69) | 12.89 (7.42)
Statistical Analysis 1: Comparison: Treatment as Usual Plus UP CBT vs Treatment as Usual; Scores on the HAM-D were analyzed using a mixed-effects linear regression analysis over 6 timepoints; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis

3. Secondary Outcome: Treatment Acceptability as Measured by Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire (CSQ) is an 8-item scale that assesses perceptions of acceptability and quality of outpatient treatment. Ratings are made on a 1 (poor) to 4 (excellent) scale for each item and then summed for a total score, with a minimum score of 8 and a maximum score of 32. Higher scores indicate greater satisfaction with treatment.
Time Frame: Six months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
Units on scale
  Baseline | 28.5 (3.79) | 27.25 (3.82)
  Month 2 | 29.43 (2.64) | 26.64 (4.40)
  Month 3 | 29.63 (3.35) | 26.22 (2.28)
  Month 4 | 28 (4.08) | 26.9 (4.28)
  Month 5 | 29.43 (3.46) | 26.6 (4.40)
  Month 6 | 29.75 (3.41) | 26.88 (4.02)
Statistical Analysis 1: Comparison: Treatment as Usual Plus UP CBT vs Treatment as Usual; Scores on the CSQ were analyzed using a mixed-effects linear regression analysis over 6 timepoints; Test type: Superiority or Other; p = 0.24, Mixed Models Analysis

4. Secondary Outcome: Association Between Anxiety Symptom Change (HAM-A) and Difficulties in Emotion Regulation Scale (DERS)
Description: Emotion regulation skills were assessed using a measure of emotion regulation (Difficulties in Emotion Regulation Scale- DERS), a 36-item Likert-type scale (1-6) calculated by averaging scores across all items. See Baseline Characteristics for baseline DERS score. See Primary Outcome Measure for a description of HAM-A.
Time Frame: Six Months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta coefficients
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
beta coefficients | .759 (.784) | .180 (1.754)
Statistical Analysis 1: Comparison: Treatment as Usual; Linear regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline DERS scores; Test type: Other; p = .62, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual Plus UP CBT; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline DERS scores; Test type: Other; p = .03, Regression, Linear

5. Secondary Outcome: Association Between Anxiety Symptom Change (HAM-A) and Reaction to Emotions (Affective Control Scale-ACS)
Description: Reactions to emotions, were assessed using the Affective Control Scale, or ACS, a 42-item Likert-type scale (1-7) calculated by averaging scores across all items. See Baseline Characteristics for baseline ACS score. See Primary Outcome Measure for description of HAM-A.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta coefficients
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
beta coefficients | .766 (.774) | .022 (1.782)
Statistical Analysis 1: Comparison: Treatment as Usual; Linear regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline ACS scores; Test type: Other; p = 0.95, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual Plus UP CBT; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline ACS scores; Test type: Other; p = 0.03, Regression, Linear

6. Secondary Outcome: Association Between Anxiety Symptom Change (HAM-A) and Anxiety Sensitivity (Anxiety Sensitivity Index-ASI)
Description: Anxiety sensitivity, were assessed using the Anxiety Sensitivity Index, or ASI, a 16-item Likert-type scale (0-4) calculated by summing scores across items. See Baseline Characteristics for baseline ASI scores. See Primary Outcome Measures for a description of HAM-A.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta coefficients
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
beta coefficients | 0.371 (1.118) | 0.062 (1.779)
Statistical Analysis 1: Comparison: Treatment as Usual; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline ASI scores; Test type: Other; p = 0.87, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual Plus UP CBT; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline ASI scores; Test type: Other; p = 0.37, Regression, Linear

7. Secondary Outcome: Association Between Anxiety Symptom Change (HAM-A) and Neuroticism (NEO Five-Factor Inventory- NEO-FFI-N)
Description: Neuroticism was assessed using the NEO Five Factor Inventory (NEO-FFI-N) which is a subscale of the NEO-FFI, a 60-item Likert-type scale (1-5) calculated by summing scores for each subscale. Only the 15-item Neuroticism subscale is included in this study. See Baseline Characteristics for baseline NEO-FFI-N. See Primary Outcome Measure for description of HAM-A.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: beta coefficients
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 13 | 15
beta coefficients | 0.720 (0.836) | 0.471 (1.572)
Statistical Analysis 1: Comparison: Treatment as Usual; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline NEO- Neuroticism scores; Test type: Other; p = 0.17, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual Plus UP CBT; Linear Regression - Dependent variable: HAM-A symptom change; Independent variable: Baseline NEO-Neuroticism scores; Test type: Other; p = .04, Regression, Linear

8. Other Pre Specified Outcome: Association Between Change on Depression (HAM-D) and Baseline Resting State Functional Connectivity of Anterior Insula and Ventrolateral Prefrontal Cortex
Description: Resting state functional magnetic resonance imaging (rsfMRI) data (non-task, eyes opened) was acquired to investigate anterior insula and ventrolateral prefrontal cortex functional connectivity as a predictor of change on depression (HAM-D). See primary outcome description of HAM-D.
Time Frame: Six Months
Population: Participating in the fMRI portion of the study was optional. A total of 15 participants consented to participate in fMRI portion (7 TAU+UP, 8 TAU). Data from all 15 subjects were analyzed.
Measure: Mean (Standard Error); unit: beta coefficient
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Number analyzed (Participants) | 7 | 8
beta coefficient | -.89 (.257) | .57 (.841)
Statistical Analysis 1: Comparison: Treatment as Usual Plus UP CBT; Fisher's z-transformed values for functional connectivity between anterior insula and ventrolateral prefrontal cortex were entered in separate treatment group-specific linear regression models as the independent variable with change in primary outcomes (HAM-D) as dependent variable; Test type: Other; p = 0.007, Regression, Linear
Statistical Analysis 2: Comparison: Treatment as Usual; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = .14, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Treatment as Usual Plus UP CBT | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual Plus UP CBT (N=13) | Treatment as Usual (N=16)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No